CLINICAL TRIAL: NCT05312346
Title: University Hospital
Brief Title: Factors Predicting Erythropoietin Responsiveness in Children on Hemodialysis at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hanan Nagdy Fawzy, pediatric specialist, Sohag University
Other Study IDs: Soh-Med-22-03-04
Record Dates: First submitted 2022-03-14; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Pediatric Patients on Hemodialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- responsiveness to erythropoietin stimulating agent: we evolute responsiveness of patients on hemodialysis for erythropoietin stimulating agents or not and factors effecting this response
  Interventions: Diagnostic Test: seum zinic,vit B12, parathyriod function

INTERVENTIONS:
Diagnostic Test: seum zinic,vit B12, parathyriod function — seum zinic,vit B12, parathyriod function

SUMMARY:
Anemia is common in patients on hemodialysis (HD) due to lack of erythropoietin (EPO) synthesis and iron deficiency is occurring in HD patients due to chronic blood loss through the dialysis circuit, repeated blood sampling, shortened red blood cell life span and lack of adherence to treatment .

Anemia is one of the most important complications that affects morbidity and mortality in chronic kidney disease (CKD) patients. It has significant impacts on those patients such as fatigue, weakness, shortness of breath, decreased quality of life, exercise capacity and physical activity, growth retardation and decreased cognitive functions, left ventricular hypertrophy, and congestive heart failure So, proper management of anemia is very important .

ELIGIBILITY:
Inclusion Criteria:

* (1) patients started dialysis in the age range of 1-18years. (2) Patient will be on regular hemodialysis.

Exclusion Criteria:

* Children who have no other co existent hematological disorder .

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: These children are attending in our Pediatric dialysis unit at Sohag University Hospital, Egypt between April 2022 and April 2023.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Hb g/dl | one year
  measure hemoglobin level
Iron profile | one year
  measure iron profile on blood
Serum creatinine | one year
  serum creatinine

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Allali S, Brousse V, Sacri AS, Chalumeau M, de Montalembert M. Anemia in children: prevalence, causes, diagnostic work-up, and long-term consequences. Expert Rev Hematol. 2017 Nov;10(11):1023-1028. doi: 10.1080/17474086.2017.1354696. Epub 2017 Oct 12. PMID 29023171
- [Background] Mikhail A, Brown C, Williams JA, Mathrani V, Shrivastava R, Evans J, Isaac H, Bhandari S. Renal association clinical practice guideline on Anaemia of Chronic Kidney Disease. BMC Nephrol. 2017 Nov 30;18(1):345. doi: 10.1186/s12882-017-0688-1. PMID 29191165
- [Background] Bamgbola OF. Pattern of resistance to erythropoietin-stimulating agents in chronic kidney disease. Kidney Int. 2011 Sep;80(5):464-74. doi: 10.1038/ki.2011.179. Epub 2011 Jun 22. PMID 21697809
- [Background] Akbari A, Clase CM, Acott P, Battistella M, Bello A, Feltmate P, Grill A, Karsanji M, Komenda P, Madore F, Manns BJ, Mahdavi S, Mustafa RA, Smyth A, Welcher ES. Canadian Society of Nephrology commentary on the KDIGO clinical practice guideline for CKD evaluation and management. Am J Kidney Dis. 2015 Feb;65(2):177-205. doi: 10.1053/j.ajkd.2014.10.013. Epub 2014 Nov 4. PMID 25511161